CLINICAL TRIAL: NCT05807256
Title: Assessment of Maternal-fetal Outcome in Pregnancy From Medically Assisted Fertilization Techniques in Women With Systemic Immunoreumatologic Diseases
Brief Title: Medically Assisted Fertilization Techniques in Systemic Immunoreumatologic Diseases
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Rovere Querini Patrizia, Associate Professor of Internal Medicine, Vita-Salute San Raffaele University Head physician, U.O. General Medicine and Continuity of Care, IRCCS San Raffaele Hospital, IRCCS San Raffaele
Other Study IDs: PMA_AD
Record Dates: First submitted 2023-03-15; First posted 2023-04-11 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Rheumatic Diseases; Fertility Disorders; Pregnancy, High Risk; Pregnancy Complications; Immunologic Disease
MeSH Terms: conditions — Rheumatic Diseases; Pregnancy Complications; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pregnant patients with systemic rheumatological diseases: pregnant patients with systemic rheumatological diseases undergoing assisted fertilization techniques
  Interventions: Other: collection and analysis of treatments and procedures already performed by normal clinical practice

INTERVENTIONS:
Other: collection and analysis of treatments and procedures already performed by normal clinical practice — The patients' anthropometric variables; laboratory test results; PMA techniques (types of fertilization/drugs used for stimulation) and the outcome of the eventual pregnancy (ongoing treatment during the pregnancy itself, development of maternal/fetal complications, such as hypertension, preeclmpsia, thrombotic events, renal failure, disease flare, neonatal outcome) and data on the type of ovarian stimulation drug treatment.

SUMMARY:
Systemic rheumatological diseases often occur in young women of childbearing age and can therefore impact fertility. There are diseases, such as arthritis, which present no contraindication to assisted reproductive techniques (ARTs), because there is no influence on the disease itself if the disease activity at conception is stable. On the other hand, patients suffering from connective tissue diseases, primarily Systemic Lupus Erythematosus (SLE) and patients suffering from primary or SLE-related Anti-Phospholipid Antibody Syndrome (APS), deserve more targeted therapies both in the context of ARTs and in the ensuing pregnancy.

To evaluate the response to ARTs in patients with systemic rheumatological diseases, both in terms of reactivation of the underlying pathology and in terms of ARTs outcome.

DETAILED DESCRIPTION:
According to standard clinical practice related to medically assisted procreation treatments, for controlled ovarian stimulation aimed at oocyte recovery, patients underwent therapy with recombinant, biosimilar, or purified human gonadotropins and eventual suppression of spontaneous ovulation with gonadotropin-releasing hormone stimulating antagonist (gnRH-antagonist), and this information will therefore be recorded. The subsequent final induction of oocyte maturity can be by purified human chorionic gonadotropin (hCG), by gonadotropin-releasing hormone stimulating hormone analog (GnRHa), or by the combination of the two, and this information will therefore also be recorded. Similarly, therapies routinely administered for endometrial preparation and luteal support during embryo transfer procedures will also be recorded (transdermal estradiol, oral estradiol; transvaginal micronized progesterone; subcutaneous progesterone). With regard to the types of PMA used, patients may have undergone homologous or heterologous procedures based on the patient's own choice and specialist indications. The IVF technique is an in vitro fertilization that consists of the union of the egg with the sperm in the laboratory -in vitro- for the purpose of obtaining already fertilized embryos to be transferred into the maternal uterus. The ICSI technique consists of intracytoplasmic sperm injection and involves the insemination of an oocyte by micro-injection of a single sperm directly into it.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with systemic immunoreumatologic disease such as SLE, APS, RA, SpA, SclS, SS, PM-DM, vasculitis
* patients who have performed one or more PMAs between January 2000 and April 2021
* patients who had their last follow-up by February 2022

Exclusion Criteria:

* Patients diagnosed with only one organ autoimmunity (e.g., diabetes mellitus I, thyroiditis of Hashimoto's, celiac disease or chronic inflammatory bowel disease in the absence of systemic disease associated);
* patients with severe renal failure, significant pulmonary hypertension or cardiomyopathy severe.

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Approximately 500 women with a definite diagnosis of systemic immunoreumatologic disease according to the criteria classificatory in place in normal clinical practice who underwent one or more PMAs between January 2000 and April 2021 will be enrolled from all participating centers.
  Pathologies examined will be:
  APS defined according to Sapporo criteria, SLE, AR, SpA, SScl, SS, PM-DM, systemic vasculitis of large- and small-medium caliber defined according to EULAR/ACR criteria.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
To quantify the risk of flare-ups of underlying immunoreumatologic disease and possible occurrence of complications during the procedure or during PMA pregnancies. | Within six months after the end of the study
  Disease flare-up will be assessed by measuring clinical parameters and antibody values ANA, ENA, SSA_SSB, antiDNA (U.A.), PMA, post PMA, post pregnancy complement.
  Complications will be evaluated in terms of maternal/fetal outcome such as hypertension, preeclmpsia, thrombotic events, renal failure, disease flare during pregnancy.
To quantify the risk of flare-ups of underlying immunoreumatologic disease and possible occurrence of complications during the procedure or during PMA pregnancies. | Within six months after the end of the study
  Disease flare-up will be assessed by measuring clinical parameters and antibody values, MB2GPI, GB2GPI (UA/mL), PMA, post PMA, post pregnancy complement.
  Complications will be evaluated in terms of maternal/fetal outcome such as hypertension, preeclmpsia, thrombotic events, renal failure, disease flare during pregnancy.
To quantify the risk of flare-ups of underlying immunoreumatologic disease and possible occurrence of complications during the procedure or during PMA pregnancies. | Within six months after the end of the study
  Disease flare-up will be assessed by measuring clinical parameters and antibody values, LAC (Microun./mL), PMA, post PMA, post pregnancy complement.
  Complications will be evaluated in terms of maternal/fetal outcome such as hypertension, preeclmpsia, thrombotic events, renal failure, disease flare during pregnancy.
To quantify the risk of flare-ups of underlying immunoreumatologic disease and possible occurrence of complications during the procedure or during PMA pregnancies. | Within six months after the end of the study
  Disease flare-up will be assessed by measuring clinical parameters and antibody values MACA, GACA, (GPL/MPL/APL unità) PMA, post PMA, post pregnancy complement.
  Complications will be evaluated in terms of maternal/fetal outcome such as hypertension, preeclmpsia, thrombotic events, renal failure, disease flare during pregnancy.

CONTACTS AND LOCATIONS:
Overall Officials: Patrizia Rovere Querini, PhD, MD, Principal Investigator — IRCCS Ospedale San Raffaele
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided